CLINICAL TRIAL: NCT00002390
Title: A Phase II Randomized, Blinded, Dose-Ranging Multicenter Study to Evaluate the Safety and Efficacy of Different Regimens of 1592U89 Monotherapy Upon Selected Immunological and Virological Markers of HIV-1 Infection in Antiretroviral Therapy-Naive Patients
Brief Title: A Study of the Safety and Effectiveness of Different Doses of 1592U89 in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 238H; CNAB2002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see if giving 1592U89 to HIV-infected patients is safe and effective in lowering viral load (level of HIV in the blood) and raising the level of CD4 cells (cells of the body that help fight infection).

DETAILED DESCRIPTION:
Patients are randomized to receive one of three doses of 1592U89. During this randomized dosing phase, if a patient meets one of the following criteria, he/she is offered open-label 1592U89 (300 mg) plus zidovudine (ZDV) plus lamivudine (3TC) (or other licensed antiretrovirals according to standard practice). Criteria are based on falling CD4 counts (return to baseline on two occasions at least 1 month apart), disease progression (defined as occurrence of a new AIDS-defining event according to CDC classification excluding CD4 counts less than 200 cells/mm3), or lack of virus suppression (defined as less than 0.7log10 reduction in viral load at Week 4 with a repeat value 1 week later, more than 5000 copies/ml HIV RNA at Weeks 12, 16, 20, or 24, or 5000 copies/ml or more anytime after Week 24).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- France (4):
  - Group Hospier Pitie-Salpetriere / Maladies Infec et Trop, Paris
  - Groupe Hospitalier Bichat-Claude Bernard, Paris
  - Hopital de Purpan / CHU de Rangueil / Medecine Interue, Toulouse
  - Hopital de Purpan / Service du Professeur Auvergnat, Toulouse
- Germany (2):
  - Universitat Erlangen, Erlangen
  - Universitatsklinikurn Frankfurt, Frankfurt

REFERENCES:
- [Background] Staszewski S, Katlama C, Harrer T, Massip P, Yeni P, Cutrell A, Tortell SM, Harrigan RP, Steel H, Lanier RE, Pearce G. A dose-ranging study to evaluate the safety and efficacy of abacavir alone or in combination with zidovudine and lamivudine in antiretroviral treatment-naive subjects. AIDS. 1998 Nov 12;12(16):F197-202. doi: 10.1097/00002030-199816000-00001. PMID 9833847